CLINICAL TRIAL: NCT02330263
Title: Effect of Preoperative Oral Carbohydrates on Postoperative Insulin Resistance in Patients Undergoing OPCAB(Off- Pump Coronary Artery Bypass Surgery)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4-2014-0908
Record Dates: First submitted 2014-12-29; First posted 2015-01-01 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Coronary Artery Occlusive Dissease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- carbohydrate group (Experimental): Randomly selected patients of the carbohydrate group are given 400ml of 12.8 g/100 ml carbohydrate beverage in the evening before their surgery and in the morning of the operation day (3 hours before their scheduled operation).
  Interventions: Dietary Supplement: carbohydrate beverage
- control group (No Intervention): Patients in the control group consume no food or drink after midnight before surgery.

INTERVENTIONS:
Dietary Supplement: carbohydrate beverage — 400ml of 12.8 g/100 ml carbohydrate beverage
  Arms: carbohydrate group

SUMMARY:
Surgical stress creates a state of insulin resistance which has been related to increased postoperative complications. Fasting before surgery induces a catabolic state that contributes to the development of insulin resistance. The aim of this study is to evaluate the effect of preoperative oral carbohydrates on postoperative insulin resistance in patients undergoing OPCAB (off-pump coronary artery bypass surgery). Sixty patients, aged 20 to 79 years, scheduled for OPCAB will be divided into carbohydrate (n=30) and control (n=30) groups. Randomly selected patients of the carbohydrate group are given 400ml of 12.8 g/100 ml carbohydrate beverage in the evening before surgery and in the morning of the operation day (3 hours before their scheduled operation). In contrast, patients in the control group consume no food or drink after midnight before their surgery. The primary endpoints are postoperative insulin resistance measured by short insulin tolerance test.

ELIGIBILITY:
Inclusion Criteria:

* patients who are scheduled to undergo OPCAB

Exclusion Criteria:

* Subjects are ineligible if they have DM(Diabetes Mellitus),
* Gastroesophageal reflux disease or gastric emptying disorder,
* inflammatory bowel disease,
* previous treatment for intra-abdominal cancer,
* entered surgery more than 5 hours after ingestion of the morning carbohydrate beverage,
* cognitive dysfunction,
* disabling mental change disorder,
* are unable to communicate or speak Korean

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2015-01; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
postoperative insulin resistance | within 1 hour after surgery

SECONDARY OUTCOMES:
preoperative discomfort | 24 hours
  the preoperative discomfort measured by VAS (Visual Analog Scale)
perioperative hemodynamic effect | 24 hours
  perioperative hemodynamic effect measured by amount of used vasopressors and minimum mixed venous oxygen saturation
postoperative complications | 24 hours
  infection, Myocardiac infarction, Acute renal failure, re-operation, death, etc

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Lee B, Soh S, Shim JK, Kim HY, Lee H, Kwak YL. Evaluation of preoperative oral carbohydrate administration on insulin resistance in off-pump coronary artery bypass patients: A randomised trial. Eur J Anaesthesiol. 2017 Nov;34(11):740-747. doi: 10.1097/EJA.0000000000000637. PMID 28437263